CLINICAL TRIAL: NCT03017989
Title: The Use of Indocyanine Green-Based Fluorescence Imaging for Intraoperative Detection of Peritoneal Endometriosis
Brief Title: ICG-Based Fluorescence Imaging for Intra-operative Detection of Endometriosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL54458.068.15
Record Dates: First submitted 2017-01-03; First posted 2017-01-11 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Endometriosis
Keywords: Near Infrared Fluorescence Imaging; Indocyanine green (ICG)
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIRF imaging (Experimental): After the white light (WL) imaging, NIRF imaging will be performed. 2.5 mg of ICG will be administered i.v. up to 5 times if needed. The lesions identified in WL, are inspected in NIRF mode. The surgeon indicated whether the lesions are more easily identified in WL or the NIRF mode and scores the visibility on a 1-10 scale. Next, inspection will take place for lesions that are seen in NIRF mode but not in WL. Biopsies will be taken from the lesions and from normal tissue for reference and sent for histology. Evaluation will take place whether the lesions differ in histological characteristics
  Interventions: Device: NIRF imaging

INTERVENTIONS:
Device: NIRF imaging — By using a fluorescence imaging device (with an adapted light source and camera), a fluorescent dye can be made visible. By injecting the fluorescent dye intravenously, the vascularization will be visible. Thereby, structures with altered vascularization are expected to 'light up' differently than the surrounding.
  Other Names: Near infrared fluorescence imaging

SUMMARY:
Endometriosis is a common disease for which the current gold standard for diagnosis is a diagnostic laparoscopy with histologic confirmation. However, during the diagnostic laparoscopy endometriotic lesions are hard to identify due to the many appearances of endometriosis. Our hypothesis is that the use of intra-operative near infrared fluorescence imaging will provide real time image enhancement for the detection of endometriotic lesions by using the different vasculature in the endometriotic lesions. This hypothesis will be tested in a prospective study with 15 patients scheduled for an elective diagnostic laparoscopy for suspected endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective laparoscopic surgery in which endometriosis is suspected
* Able to understand the nature of the study and what will be required of them
* Females
* Age >18years
* Premenopausal
* No history of impaired liver and renal function
* No history of hypersensitivity or allergy to indocyanine green or iodide
* No hyper-thyroidism or autonomic thyroid adenomas
* Willing to participate

Exclusion Criteria:

* Not able to give written informed consent
* Males
* Aged < 18 years
* Pregnant or breast-feeding women
* Known hypersensitivity or allergy to indocyanine green or iodide
* Known hyper-thyroidism or autonomic thyroid adenomas
* Not willing to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Number of detected endometriotic lesions with Near Infrared Light versus with white light | during surgery
  The number of lesions detected in near-infrared light will be compared to the number of endometriotic lesions seen in white light. Hereby, we aim to investigate whether all lesions seen in white light are also seen in NIRF light and whether NIRF light shows endometriotic lesions that were not visible in white light.

SECONDARY OUTCOMES:
Histological assessment of taken biopsies: assessment of localization of ICG uptake | biopsies taken during surgery, which are assessed during the 1th week after surgery
  Hereby, we aim to investigate whether the different histological subtypes of endometriosis light up differently in NIRF light. We interested in whether there is another localisation of ICG uptake at cellular level in the different histological subtypes.
Time measurement | during the laparoscopic procedure
  measuring the total operating time, and the extra time needed for fluorescence imaging
Safety of the procedure: assessment of complications during the procedure attributable to the technique or dye | during surgery
  Complications during the diagnostic laparoscopy attributable to the imaging technique or dye are described here.
Satisfaction of the surgeon with the technique | immediately after surgery
  Immediately the surgeon will be asked whether he/she considered the use of NIRF imaging an useful additive to the procedure.
Histological assessment of taken biopsies: assessment Target to background ratio | biopsies taken during surgery, which are assessed during the 1th week after surgery
  The biopsies taken during surgery will be analysed together with the video recordings. Hereby, we aim to investigate whether the different histological subtypes of endometriosis light up differently in NIRF light. We interested in whether there is another target to background rato in the different histological subtypes.

CONTACTS AND LOCATIONS:
Overall Officials: Laurents Stassen, M.D, Ph.D, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided